CLINICAL TRIAL: NCT04955886
Title: Efficacy and Safety of Surufatinib Combined With Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma : a Prospective, Single Arm and Multicenter Trial
Brief Title: Surufatinib Combined With Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-HNC104
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent or Metastatic Nasopharyngeal Carcinoma. (Experimental): Patients with Recurrent or Metastatic Nasopharyngeal Carcinoma were given Surufatinib Combined With Toripalimab.
  Interventions: Drug: Surufatinib(HMPL-012)

INTERVENTIONS:
Drug: Surufatinib(HMPL-012) — Surufatinib(250mg) will be orally administered within 1 hour after breakfast once a day (QD) , Toripalimab was administered intravenously at a fixed dose of 240 mg, and the infusion time was 60 ± 5 min, once every 21 days. The cumulative longest medication period is 2 years. Until disease progression, death, intolerable toxicity or other protocol specified end-of-treatment criteria is met .
  Other Names: Toripalimab

SUMMARY:
A prospective, single-arm,mutil-center study to assess the efficacy and safety of Surufatinib combined with Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma.

DETAILED DESCRIPTION:
This study adopt Simon's two-stage Optimal designs method based on the primary endpoint of objective response rates. 4 patients were planned for the first stage. If one or more responses were observed, an additional 8 patients were to be accrued for a total of 12 patients. If 4 or more of the 12 patients achieved an objective response, then this study was designated worthy of additional investigation.Considering a 10% abscission rate, a total of 14 patients were included.

Surufatinib（250mg) will be orally administered within 1 hour after breakfast once a day (QD) , Toripalimab was administered intravenously at a fixed dose of 240 mg, and the infusion time was 60 ± 5 min, once every 21 days. The cumulative longest medication period is 2 years. Until disease progression, death, intolerable toxicity or other protocol specified end-of-treatment criteria is met .

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures;
2. Male and Female aged between 18 and 75 years are eligible;
3. Histologically or cytologically confirmed that Recurrent or Metastatic Nasopharyngeal Carcinoma.
4. Patients must have received at least one standard platinum-based systemic chemotherapy regimen for the treatment of recurrent or metastatic NPC;Or the insensitivity or intolerance to platinum when the patient has previously received radical therapy;
5. Not suitable for local treatment (no radiotherapy or surgery);
6. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria;
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
8. Screening laboratory values must meet the following criteria (within past 14 days):

   * neutrophils ≥1.5×109/L ;
   * platelets ≥100×109/L；
   * hemoglobin ≥ 10 g/dL;
   * total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1.5╳ULN;
9. Ability to follow the program;
10. Toxic side effects of any previous chemotherapy have returned to less than or equal to NCI CTCAE1 level or baseline;
11. Predicted survival >3 months;
12. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. The pathological type was neuroendocrine or small cell carcinoma;
2. Evidence with active CNS disease or previous brain metastases;
3. Prior received anti-tumor monoclonal antibodies or other investigational drugs within the first 4 weeks of enrollment;Previous treatment with other anti-PD-1 antibodies or other treatments targeting PD-1 / PD-L1.
4. Prior treatment with Surufatinib,or other antiangiogenic drugs were used ;
5. Patients were on immunosuppressive or systemic hormone therapy (doses greater than 10mg/day prednisone or other equivalent hormone) for immunosuppressive purposes and were still on it within 2 weeks prior to enrolment;
6. The patient has any active autoimmune disease or a history of autoimmune disease;
7. Have clinical cardiac symptoms or diseases that are not well controlled;
8. Patients with congenital or acquired immune deficiency;
9. Chemotherapy, targeted therapy and radiotherapy were received within 2 weeks before enrollment;
10. Patients who had a history of gastrointestinal perforation or had undergone major surgery 4 weeks before enrollment;
11. During the first 6 months of enrollment, there were arterial/venous thrombosis events, such as non-cardiovascular and cerebrovascular (including temporary ischemic attack), deep vein thrombosis (except for venous thrombosis caused by intravenous catheterization during pre-chemotherapy, which was determined by the investigators to be cured), and pulmonary embolism;
12. Patients with abnormal coagulation function (International normalized ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN), bleeding tendency (such as active ulcer lesions in the stomach, occlusive blood in the stool (++), melenia and/or hematemesis and hemoptysis within 3 months) or lesions close to large vessels.The lesions involved in the skin or mucosal cavity are at risk of rupture;
13. Hypertension that cannot be controlled by medication;
14. Routine urine indicated more than 2+ urine protein or 24 hours urine protein >150mg/L;
15. Calibration of QT interval > 470MSEC;If the patient has an extended QT interval, but the investigator's study evaluates the prolonged period as due to a pacemaker (and no other cardiac abnormality), it is up to the investigator to determine whether the patient is eligible for the study;
16. Had other malignant tumors in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled);
17. Known to be allergic to drug ingredients;
18. Patients at risk of massive bleeding in the nasopharynx or deep ulcers in the nasopharynx.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib and Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma. patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  OS was calculated from the date of pharmacy to death from any cause.
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Duration of relief (DOR) | through study completion, an average of 1 year
  The length of time that a tumor continues to respond to treatment without the cancer growing or spreading.

CONTACTS AND LOCATIONS:
Overall Officials: Sufang Qiu, MD, Principal Investigator — Fujian Cancer Hospital
Locations (2):
- China (2):
  - Affiliated Cancer Hospital of Sun Yat-sen University, Guangdong
  - Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai